CLINICAL TRIAL: NCT01707745
Title: Efficacy and Safety of Intravitreal Bevacizumab for Threshold ROP.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sivakami A Pai (Other Government)
Responsible Party: Sponsor-Investigator, Sivakami A Pai, Doctor, Dubai Health Authority
Organization: Dubai Health Authority (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Avastin for threshold ROP.
Record Dates: First submitted 2012-09-22; First posted 2012-10-16 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Stage 2+ or Stage 3+ Retinopathy of Prematurity in Zone I or Zone II.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Avastin (Other): Bevacizumab(Avastin) 0.75mg in 0.03 ml
  Interventions: Procedure: Intravitreal Bevacizumab

INTERVENTIONS:
Procedure: Intravitreal Bevacizumab
  Other Names: Intravitreal Avastin

SUMMARY:
Prospective study to evaluate the efficacy and safety of intravitreal bevacizumab In retinopathy of prematurity (ROP).

Bevacizumab 0.75 mg in 0.03 ml was given to stage 2+ or stage 3+ ROP in Zone I or Zone II.

ELIGIBILITY:
Inclusion Criteria: stage 2+ or stage 3+ Retinopathy of prematurity in Zone I or Zone II.

Informed written consent by parents or guardian.

-

Exclusion Criteria:

Refusal to give consent Critically ill neonates.

-

Ages: 32 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Regression Of ROP | Minimum 6 months follow up after intravitreal Avastin

SECONDARY OUTCOMES:
Recurrence of ROP | minimum 6 months of follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Dubai Hospital, Dubai, UAE, United Arab Emirates